CLINICAL TRIAL: NCT01387685
Title: Treatment of Pelvic Organ Prolapse by PIVS Versus Surgeon Cut Mesh
Status: Withdrawn | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Dr. Menahem Neuman, Western Galilee Hospital and vaious clinics
Other Study IDs: 920090042
Record Dates: First submitted 2011-06-29; First posted 2011-07-04 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Pelvic Floor Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Women with pelvic floor prolapse who underwent surgery with mesh will be enrolled. The investigators will compare data from the chart, telephone interviews and physical examinations between those who underwent mesh placement to those who underwent placement of PIVS.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent surgery for pelvic floor prolapse

Exclusion Criteria:

* Women who did not have surgery for pelvic floor prolapse.

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who underwent surgery for pelvic floor prolapse who underwent surgery by eithe surgeon-cut-mesh or by PIVS
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with study outcome | six to twelve months after surgery

SECONDARY OUTCOMES:
Side effects of the surgery: pain, vaginal erosion by tape, bleeding | Within six to twelve months after study

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Department of Obstetrics and Gynecology, Western Galilee Hospital, Nahariya
  - Dr Neuman clinic, Tel Aviv